CLINICAL TRIAL: NCT06886919
Title: Clinical Study Evaluating the Safety and Efficacy of IC19 CAR-T Cell Therapy for Refractory Systemic Lupus Erythematosus
Acronym: IC19 CAR-T
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beijing Immunochina Medical Science & Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZMA03
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Difficult to Treat Systemic Lupus Erythematosus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with refractory systemic lupus erythematosus (Experimental): The "3+3" dose escalation method will be adopted, with 1 × 10 ^ 8 CAR-T cells/dose and 2 × 10 ^ 8 CAR-T cells/dose, and two dose groups increasing sequentially. Due to the specificity of cell preparations, it is allowed for the actual dosage of each dose group to fluctuate by ± 30%.
  Interventions: Biological: Engineering of chimeric antigen receptors targeting CD19 in allogeneic T cells

INTERVENTIONS:
Biological: Engineering of chimeric antigen receptors targeting CD19 in allogeneic T cells — About 6 subjects will be included in the study, and a "3+3" dose escalation method will be used. The dosage will be gradually increased in two dose groups: 1 × 10 ^ 8 CAR-T cells/dose and 2 × 10 ^ 8 CAR-T cells/dose. Three subjects are enrolled in each dose group first, and within the same dose group, the cell transfusion interval between the first two subjects should not be less than 14 days. If no dose limiting toxicity (DLT) is observed in a certain dose group, the dose will be increased to the next dose; If one case of DLT occurs, this dose group needs to be divided into three additional subjects (a total of six subjects). If no new DLT occurs, the dosage will be increased to the next dose; If more than 1/6 of the 6 subjects develop DLT, the dose escalation will be terminated, and the Safety Review Committee (SRC) will discuss whether to reduce the dose and continue the monotherapy study.
  Other Names: IC19 CAR-T cells

SUMMARY:
This study is an open label, single arm exploratory clinical trial of IC19 CAR-T cell therapy for refractory systemic lupus erythematosus. Patients who are still in an active state after systemic treatment using the standard treatment regimen specified in the treatment guidelines were selected to receive IC19 CAR-T cell single pulse infusion therapy.

DETAILED DESCRIPTION:
1. The "3+3" dose escalation method will be adopted, with 1 × 10 ^ 8 CAR-T cells/dose and 2 × 10 ^ 8 CAR-T cells/dose, and two dose groups increasing sequentially. Due to the specificity of cell preparations, it is allowed for the actual dosage of each dose group to fluctuate by ± 30%.
2. Three subjects are enrolled in each dose group first, and within the same dose group, the cell transfusion interval between the first two subjects should not be less than 14 days. If no dose limiting toxicity (DLT) is observed in a certain dose group, the dose will be increased to the next dose; If one case of DLT occurs, this dose group needs to be divided into three additional subjects (a total of six subjects). If no new DLT occurs, the dosage will be increased to the next dose; If more than 1/6 of the 6 subjects develop DLT, the dose escalation will be terminated, and the Safety Review Committee (SRC) will discuss whether to reduce the dose and continue the monotherapy study.
3. Definition of DLT: Any of the following events related to the investigational drug (definitely related, likely related, possibly related) that occur within 28 days after a subject receives any IC19 CAR-T cell infusion:

1) Any grade 4 or 5 adverse events related to IC19 CAR-T cells that occur after treatment, excluding laboratory test indicators of no clinical significance; 2) Any grade 3 adverse events related to IC19 CAR-T cells that occur after treatment and do not improve to ≤ grade 2 within 7 days, excluding clinically insignificant laboratory test indicators; 3) Any grade 3 epileptic seizures that occur after treatment and cannot be relieved to ≤ grade 2 within 3 days;

The following expected events will not be considered DLT:

Hematology:

1. Grade 3 neutropenia or Grade 4 neutropenia lasting no more than 28 days;
2. Grade 3 or 4 leukopenia;
3. Grade 3 or 4 lymphocyte reduction;
4. Grade 3 anemia or Grade 4 anemia lasting no more than 28 days;
5. Grade 3 thrombocytopenia or Grade 4 thrombocytopenia lasting no more than 28 days;
6. Other types of blood cell reduction besides those mentioned above.

Non hematology:

1. Grade 3 transaminase and bilirubin elevation should be restored to ≤ Grade 2 within 2 weeks;
2. Grade 3 hemophagocytic syndrome recovers to ≤ Grade 2 within 2 weeks;
3. Grade 3 chills, recover to ≤ Grade 2 within ≤ 72 hours;
4. Grade 3 hypotension (without other CRS symptoms), requiring vasopressor support and recovering to ≤ Grade 2 within ≤ 72 hours;
5. Level 3 CRS, recover to ≤ Level 2 within ≤ 72 hours;
6. Grade 3 ICANS ≤ 7 days, with remission to ≤ Grade 2 within 1 week and remission to baseline within ≤ 28 days.

For grade 3 or 4 toxicity that occurs after 28 days of IC19 CAR-T cell transfusion, SRC will discuss the specific situation. In this study, except for CRS and ICANS, which will be classified according to the ASTCT 2019 consensus grading criteria, adverse events of subjects will be classified according to the National Cancer Institute (NCI) Common Terminology for Adverse Events (CTCAE 5.0).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects diagnosed with systemic lupus erythematosus who meet the 2019 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) classification criteria for SLE;
2. Prior to screening, treatment with glucocorticoids (sufficient or shock therapy) combined with immunosuppressants (cyclophosphamide, mycophenolate mofetil, antimalarial drugs, azathioprine, methotrexate, leflunomide, tacrolimus, cyclosporine, etc.) and at least one biological agent (rituximab, belimumab, tacrolizumab, etc.) must have been received for at least 2 months, and the dosage must be stable for more than 2 weeks. The disease should still be active or recur after disease remission.

Oral corticosteroids need to meet the following conditions:

1. Prednisone (or equivalent) ≥ 7.5 mg/day and ≤ 60 mg/day;
2. When used in combination with immunosuppressants and/or biologics, there is no minimum daily dose requirement for glucocorticoids.

3. When screening, the disease activity score (SLEDAI-2000) should be ≥ 8 points; 4. During the screening period, it meets the criteria of being positive for anti nuclear antibodies (ANAs), anti dsDNA antibodies, or anti Smith antibodies.

5. Age range of 18-70 years old (including threshold), gender not limited; 6. Expected survival period of more than 3 months; 7. The functions of important organs meet the following requirements:

1. The bone marrow function needs to meet the following requirements: a. Neutrophil count ≥ 1 × 109/L; b. Platelets ≥ 50 × 109/L; c. Hemoglobin ≥ 60g/L;
2. Liver function: ALT ≤ 2.5 × ULN (upper limit of normal, ULN), AST ≤ 2.5 × ULN; TBIL ≤ 1.5 × ULN (for subjects with Gilbert syndrome, ALT and AST ≤ 5 × ULN, total bilirubin ≤ 3.0 × ULN);
3. Renal function: creatinine ≤ 1.5 × ULN or creatinine clearance rate (CrCl) ≥ 40 ml/min (Cockcroft/Gault formula);
4. Coagulation function: International normalized ratio (INR) ≤ 1.5 × ULN, prothrombin time (PT) ≤ 1.5 × ULN;
5. Cardiac function: Good hemodynamic stability, left ventricular ejection fraction (LVEF) ≥ 50%;
6. Finger pulse oxygen saturation ≥ 92% in non oxygen state; 8. Women of childbearing age who have a negative blood pregnancy test before the start of the trial and agree to participate in the trial until the last time Visit individuals who have adopted effective contraceptive measures; Male participants with reproductive partners agree to take effective contraceptive measures during the trial period until the last follow-up; And not in the lactation period.

9. The individual or legal guardian agrees to participate in this experiment and signs the informed consent form.

Exclusion Criteria:

1. Diseases of the central nervous system that have clinical significance in the past or during screening, such as seizures, epilepsy, epileptic seizures, cerebrovascular disease (ischemia/hemorrhage), cerebral edema, reversible posterior white matter encephalopathy, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, encephalitis, CNS vasculitis, or psychiatric disorders;
2. Screening for acute severe lupus nephritis within the first 2 months, defined as significant deterioration of kidney disease (such as the presence of urine sediment and other laboratory abnormalities) that the researcher believes may require the use of contraindicated drugs or high-dose corticosteroids (prednisone ≥ 100 mg/d or equivalent corticosteroid treatment ≥ 14 days) for treatment in the first 2 months of the study.
3. If there is an uncontrolled lupus crisis within the first 2 months of screening, the researcher has assessed that it is not suitable to participate in this study;
4. A large amount of serous fluid accumulation (such as pleural effusion and peritoneal effusion) with compression symptoms that cannot be controlled after treatment;
5. Other active autoimmune diseases (such as Crohn's disease and rheumatoid arthritis) that require systemic immunosuppressive therapy within the first 2 years of screening, except for SLE;
6. Patients who have received or are waiting for hematopoietic stem cell/bone marrow transplantation or organ transplantation in the past;
7. Individuals who have previously received gene modified cell therapy, such as TCR-T therapy, CAR-T therapy, etc;
8. Screening for clinical study drugs used for any other autoimmune diseases within the first 3 months. But if the research treatment is ineffective or if the disease progresses, and at least 5 half lives have passed before screening, it is allowed to be included in the group;
9. Have a history of ≥ grade 2 bleeding within 30 days prior to screening, or require long-term continuous use of anticoagulant drugs (such as warfarin, low molecular weight heparin, or Xa factor inhibitors) for treatment;
10. Vaccination with live or attenuated vaccines within 6 weeks prior to screening;
11. Active hepatitis B or hepatitis C virus is defined as: subjects who are positive for hepatitis B B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and whose peripheral blood HBV-DNA detection is higher than the lower limit of detection (HBsAg positive but whose peripheral blood HBV-DNA detection is lower than the lower limit of detection according to the Guidelines for the Prevention and Treatment of Chronic Hepatitis B, Version 2022, at least 4 weeks of antiviral treatment shall be carried out before the first use of the study drug, and antiviral treatment shall be continued for 6-12 months during the study process, and the levels of HBV-DNA, HBsAg and ALT shall be monitored every 1-3 months); Hepatitis C virus (HCV) antibody positive and peripheral blood HCV-RNA detection above the detection limit; HIV antibody positive; Positive syphilis antibody;
12. Active EB virus and cytomegalovirus, defined as: subjects with positive or negative IgM antibodies in EB virus serum but EBV-DNA higher than normal values; Subjects with IgM antibody positive or IgM antibody negative but CMV-DNA higher than normal in the serum of cytomegalovirus (CMV);
13. Within the past year, there have been severe chronic obstructive pulmonary disease, interstitial lung disease, severe asthma, and clinically significant abnormalities in lung function tests, such as moderate to severe pulmonary arterial hypertension (average pulmonary arterial pressure detected by echocardiography>60mmHg) that require oxygen storage mask oxygen therapy or non-invasive or invasive ventilator assisted breathing during screening; Interstitial lung disease related to autoimmune diseases must meet all inclusion criteria;
14. Hypertension with poor drug control (systolic blood pressure>160mmHg and/or diastolic blood pressure>90mmHg) or a history of any of the following cardiovascular diseases within 6 months prior to screening: long QTc syndrome or QTc interval>480 ms; Complete left bundle branch block, grade II/III atrioventricular block; Severe and uncontrolled arrhythmias requiring medication treatment; History of chronic congestive heart failure and NYHA ≥ 3 (refer to Appendix 2) with a heart ejection fraction below 50% within the 6 months prior to screening; Heart valve disease with CTCAE ≥ 3 grade; Within the first 6 months of screening, there has been a history of myocardial infarction, cardiac angioplasty or stent implantation, unstable angina, severe pericardial disease, or other clinically significant heart diseases;
15. History of symptomatic deep vein thrombosis or pulmonary embolism within the past 6 months prior to the start of screening;
16. Other untreated malignant tumors within the past 5 years or simultaneously, excluding cervical cancer in situ, basal cell carcinoma of the skin, and ductal carcinoma in situ of the breast;
17. Infections (fungi, bacteria, viruses, or others) that require intravenous injection of antibiotics for control or are uncontrollable For simple urinary tract infections and bacterial pharyngitis, if the researchers evaluate that they can be controlled through treatment, they can be included in the study;
18. Individuals who are known to have allergic reactions, hypersensitivity reactions, intolerance, or contraindications to any ingredients of drugs that may be used in the study (including fludarabine, cyclophosphamide, tocilizumab, albumin), or who have previously experienced severe allergic reactions;
19. Have a history of alcohol or drug abuse in the past 24 weeks;
20. The researcher shall determine whether the subjects have any factors that affect compliance with the protocol, or are unwilling or unable to comply with the procedures required in the research protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of IC19 CAR-T cell therapy for refractory systemic lupus erythematosus | 28 days after IC19 CAR-T cell transfusion
  The incidence of adverse events related to IC19 CAR-T cell transfusion within 28 days after IC19 CAR-T cell transfusion, abnormal laboratory test results with clinical significance, including dose limited toxicity (DLT).

SECONDARY OUTCOMES:
Evaluate the efficacy of IC19 CAR-T cell therapy in the treatment of refractory systemic lupus erythematosus | 24 weeks after IC19 CAR-T cell reinfusion
  Changes in SLE Disease Activity Index (SLEDAI-2K) scores (0-105 points; 0-4 points: almost no activity; 5-9 points: mild activity; 10-14 points: moderate activity; ≥ 15 points: severe activity) compared to baseline at 12 and 24 weeks after IC19 CAR-T cell transfusion
Evaluate the efficacy of IC19 CAR-T cell therapy in the treatment of refractory systemic lupus erythematosus | 24 weeks after IC19 CAR-T cell reinfusion
  Changes in the British Islet Lupus Assessment Group Index (BILAG-2004) compared to baseline at 12 and 24 weeks after IC19 CAR-T cell reinfusion
Evaluate the efficacy of IC19 CAR-T cell therapy in the treatment of refractory systemic lupus erythematosus | 24 weeks after IC19 CAR-T cell reinfusion
  The overall assessment (PGA) of clinical physicians at 12 and 24 weeks after IC19 CAR-T cell reinfusion compared to baseline changes
Evaluate the efficacy of IC19 CAR-T cell therapy in the treatment of refractory systemic lupus erythematosus | 24 weeks after IC19 CAR-T cell reinfusion
  The proportion of subjects who reached SLE response index 4 (SRI-4) at 12 and 24 weeks after IC19 CAR-T cell reinfusion
Evaluate the efficacy of IC19 CAR-T cell therapy in the treatment of refractory systemic lupus erythematosus | 24 weeks after IC19 CAR-T cell reinfusion
  The proportion of subjects who reached lupus low disease activity state (LLDAS) at 12 and 24 weeks after IC19 CAR-T cell reinfusion
Evaluate the efficacy of IC19 CAR-T cell therapy in the treatment of refractory systemic lupus erythematosus | 24 weeks after IC19 CAR-T cell reinfusion
  Proportion of subjects who achieved disease remission (DORIS) after IC19 CAR-T cell transfusion at 12 and 24 weeks
Evaluate the efficacy of IC19 CAR-T cell therapy in the treatment of refractory systemic lupus erythematosus | 24 weeks after IC19 CAR-T cell reinfusion
  Changes in Systemic Lupus Erythematosus Disease Activity Score (SLE-DAS) from baseline at 12 and 24 weeks after IC19 CAR-T cell reinfusion
Evaluate the efficacy of IC19 CAR-T cell therapy in the treatment of refractory systemic lupus erythematosus | 48 weeks after IC19 CAR-T cell transfusion
  The changes in various indicators from baseline at other time points after IC19 CAR-T cell transfusion, such as weeks 4, 8, 16, 20, 36, and 48, as mentioned in items 1-7 above
Evaluate the efficacy of IC19 CAR-T cell therapy in the treatment of refractory systemic lupus erythematosus | 48 weeks after IC19 CAR-T cell transfusion
  Changes in quality of life (SF-36) compared to baseline at 12, 24, and 48 weeks after IC19 CAR-T cell transfusion
Evaluate the pharmacokinetic (PK) and pharmacodynamic (PD) characteristics of IC19 CAR-T cell therapy for refractory systemic lupus erythematosus | 48 weeks after IC19 CAR-T cell transfusion
  Changes in immunoglobulin (IgG, IgM, IgA, IgE), antibody (anti ds DNA antibody, anti nuclear antibody ANA), and complement (C3, C4) levels after IC19 CAR-T cell transfusion
Evaluate the pharmacokinetic (PK) and pharmacodynamic (PD) characteristics of IC19 CAR-T cell therapy for refractory systemic lupus erythematosus | 48 weeks after IC19 CAR-T cell transfusion
  After IC19 CAR-T cell transfusion, the peak time (Tmax), amplification peak (Cmax), area under the curve (AUC), and retention time of CAR-T cells in the patient's peripheral blood
Evaluate the pharmacokinetic (PK) and pharmacodynamic (PD) characteristics of IC19 CAR-T cell therapy for refractory systemic lupus erythematosus | 48 weeks after IC19 CAR-T cell transfusion
  Changes in CD19+B cell levels and major B cell functional subgroups (initial B cells, memory B cells, category switching B cells) in peripheral blood after IC19 CAR-T cell transfusion
Evaluate the pharmacokinetic (PK) and pharmacodynamic (PD) characteristics of IC19 CAR-T cell therapy for refractory systemic lupus erythematosus | 48 weeks after IC19 CAR-T cell transfusion
  The level of anti drug antibodies (ADA) after IC19 CAR-T cell reinfusion

CONTACTS AND LOCATIONS:
Overall Officials: yajing Zhang, doctorate, Principal Investigator — Beijing Gaobo Boren Hospital

IPD SHARING:
Plan to Share IPD: No